CLINICAL TRIAL: NCT06986070
Title: A Phase 1, First-in-Human, Clinical Trial to Evaluate the Safety of Small Mobile Stem Cells (SMS) Delivered Into the Lung as a Potential Organ Regeneration Therapy in Chronic Obstructive Pulmonary Disease (SORT-COPD Study
Brief Title: Investigation of Small Mobile Stem Cells (SMS Cells) in Participants With Chronic Obstructive Pulmonary Disease (COPD).
Acronym: SORT-COPD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SMSbiotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A005; ACTRN12624001140549 (Registry Identifier: Australia New Zealand Clinical Trial Registry (ANZCTR))
Record Dates: First submitted 2025-03-13; First posted 2025-05-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spermine Synthase; Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants in the cohort 1 (low dose) will receive 1.2 billion cells/ml. (Experimental): Dose escalating Cohort 1.
  Interventions: Biological: Stem cells
- Participants in the cohort 2 (medium dose) will receive 2.4 billion cells/ml. (Experimental): Dose escalating Cohort 2.
  Interventions: Biological: Stem cells
- Participants in the cohort 3 (high dose) will receive 4.8 billion cells/m (Experimental): Dose Escalating Cohort 3.
  Interventions: Biological: Stem cells

INTERVENTIONS:
Biological: Stem cells — The suspension of stem cells will be put in a medical nebulizer machine, commonly used to deliver medicines into the lungs through inhalation. This means that the participants will breathe in the mist containing the SMS cells, produced by the nebulizer machine. This is a Phase I First-in-Human study, which indicates that this treatment is being studied for the first time in humans.
  Other Names: Small Molecule Stem (SMS) Cells

SUMMARY:
This study is a phase 1, first-in-human, open-label, non-randomized, dose escalation safety study of 18 participants, between 39 and 69 years of age, with mild to moderate chronic obstructive pulmonary disease, treated with SORT-COPD (SMS cells).

The primary objective of this study is to determine the safety of SORT-COPD (SMS cells) at three doses in people with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
The suspension of stem cells will be put in a medical nebulizer machine, commonly used to deliver medicines into the lungs through inhalation. This means that the participants will breathe in the mist containing the SMS cells, produced by the nebulizer machine. This is a Phase I First-in-Human study, which indicates that this treatment is being studied for the first time in humans.

18 participants are expected to be enrolled into this study. Participants will be divided into three groups of six volunteers, with the first group receiving the lowest dose of the study treatment, the second group receiving a higher dose, and the third group receiving the highest dose. Between each of the three groups, there will be a pause to permit detection of any short-term adverse effects of the treatment at a specific dose.

Participants will be treated with the study drug, SORT COPD (Small Mobile Stem Cells), delivered via a medical nebuliser on the 1st, 4th, and the 8th days of the study in-clinic. The nebuliser treatment involves inhaling mist from a mouthpiece attached to a standard medical nebuliser machine and takes about 10 to 15 minutes to complete.

The volume to be nebulised is 3 millilitres (less than one teaspoon). Participants in the cohort 1 (low dose) will receive 1.2 billion cells/ml. Participants in the cohort 2 (medium dose) will receive 2.4 billion cells/ml. Participants in the cohort 3 (high dose) will receive 4.8 billion cells/ml.

The study treatment (SMS) cells will be given in three different concentrations with the lowest dose given to the 1st group of 6 participants, with the dose doubled for each group. The members of each group will receive the same dose at each treatment visit.

Participants will actively be in the study for up to 5 or 6 weeks, including the initial screening and testing period before the treatment is applied, during treatment, and about 4 weeks after the first treatment. Also, about 3 to 6 months after the study, participants will be contacted via telephone to answer some questions about their state of health, which will be the end of the study.

Individual participant duration will be up to a maximum of 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 39 to 69 years (inclusive).
2. Female participants:

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

   Is a woman of nonchildbearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method from screening until 30 days after the last dose of study intervention.

   A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) at Screening and on Day 1, prior to administration of study intervention.

   If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

   The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
3. Male participants:

   Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 30 days after the last dose of study intervention:

   Refrain from donating fresh unwashed semen. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR must agree to use contraception/barrier (male condom).
4. Has a diagnosis of mild or moderate COPD-C (cigarette smoking COPD) or COPD-P (biomass and pollution exposure COPD) according to the 2023 Global Initiative for Chronic Obstructive Lung Disease (GOLD) Criteria.

   Lung impairment will be determined with post-bronchodilator FEV1 spirometry.
5. Has previously received treatment for COPD-C or COPD-P.
6. Has stable COPD disease state, defined as no exacerbations in the 12 weeks prior to screening, no hospitalizations in the 12 weeks prior to screening, and no changes in COPD medication in the 28 days prior to screening.
7. Agrees to comply with study specific procedures and visits, including non-smoking during the treatment and follow-up periods of the study.
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Previous or current diagnosis of COPD-G, COPD-D, COPD-I, COPD-A or COPD-U; asthma, congestive heart failure, bronchiectasis, tuberculosis, obliterative bronchiolitis or diffuse panbronchiolitis.
2. Previous or current history of respiratory failure other than due to COPD (e.g. restrictive lung disease, sarcoidosis, tuberculosis, idiopathic pulmonary fibrosis, bronchiectasis, CMV pneumonitis, cystic fibrosis, asbestosis, silicosis or farmer's lung disease), or detection of any of these conditions through screening CT scanning.
3. History of COVID associated pneumonia with hypoxemic respiratory failure in the 12 weeks prior to screening.
4. Current use, or use within 21 days of screening, of systemic corticosteroids. Participants on inhaled corticosteroids or combined inhaled therapies can be included, however must schedule inhaled therapies 12 hours prior to dosing IP and 12-hours post dosing IP.
5. Any history of chronic liver disease, or abnormal liver function at screening, defined as:

   Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) more than 2.5 times the upper limit of normal (ULN) Total bilirubin more than two times the ULN Participants with documented Gilbert's syndrome are permitted to enter the study.
6. History of chronic renal insufficiency, defined as and eGFR < 90 mL/min/1.73 m2. Participants without a history of chronic renal insufficiency, who at screening have an eGFR detected between 60-89 mL/min/1.73 m2, should have their eGFR repeated as per standard clinical procedure.
7. Uncontrolled hypertension, or current hypertension controlled on more than two medications.
8. History, within the last two years, of coronary artery disease, coronary artery bypass graft surgery, percutaneous transluminal coronary angioplasty, severe peripheral arterial disease, cerebrovascular disease (including history of transient ischemic attack or cerebrovascular accident), or any such history that, in the opinion of the investigator, will impact participation in the study.
9. Type 1 or Type 2 diabetes mellitus with glycosylated hemoglobin (HbA1c > 7.5%) at screening.
10. No active malignancy in the last three years, including any potential neoplasm detected via high-resolution CT scan (nodule > 5 mm) detected as part of the screening process.

    People with a history of basal cell or squamous cell carcinoma of the skin are eligible.
11. History of HIV or other immunosuppressed conditions, Hepatitis B or Hepatitis C, or use of immunosuppressive medications within 14 days prior to screening, and for 3 weeks after the last dose of study intervention is administered.
12. Active infection requiring systemic antibiotic treatment within 12 weeks prior to screening.
13. Body mass index (BMI) > 60 kg/m2.
14. Active smoking of tobacco, cannabis or vaping in the 28 days prior to screening as indicated by results of cotinine urine testing, performed at screening. Use of nicotine containing products such as nicotine patches, oral nicotine products or nicotine chewing gum is permitted, noting that cotinine results will be positive. Positive results will be documented by the investigator as "attributed to permitted nicotine products".
15. History of alcohol or other substance abuse, with sobriety less than one year, or that in the opinion of the investigator, will impact participation in the study.
16. Pregnant or breastfeeding.
17. Any severe medication allergy, including an allergy to bovine products.
18. Any other medical condition, psychiatric condition or illness, that according to the Principal Investigator might render the subject unlikely to tolerate the inhalation of SORT-COPD (SMS cells), or to complete the study.
19. Current participation in any other clinical trial or participation in the last six weeks or subject received an experimental therapy (drug or biologic) for any indication within 12 months prior to enrolment.
20. Unable or unwilling to comply with study specific schedules or procedures.

Ages: 39 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events. | Day 1, 2, 3, 4, 5, 8, 9, 21, 28, Month 3 and Month 6.
  Treatment emergent adverse events and serious adverse events.
Dose limiting toxicity. | Day 1, 2, 3, 4, 5, 8, 9, 21, 28, Month 3 and Month 6.
  Any treatment emergent adverse event that ii treatment related and classified as severe or the event is classified as a serious adverse event.
Safety laboratory testing | Screening, Day 2, 3, 5, 9, 21 and 28.
  All laboratory parameters will be summarized using descriptive statistics for each cohort and overall, for all time points assessed, including change from baseline for all post-dose assessments. Selected laboratory test results will be graded in accordance with the NCI CTCAE criteria.

SECONDARY OUTCOMES:
Spirometry | Screening, Day 1, 2, 3, 4, 5, 8, 9, 21 and 28.
  To be performed according to the American Thoracic Society/European Respiratory Society Standards. Forced Expiratory Volume in 1 second (FEV1) measured in liters (L).
Spirometry | Screening, Day 1, 2, 3, 4, 5, 8, 9, 21 and 28.
  To be performed according to the American Thoracic Society/European Respiratory Society Standards. Forced Vital Capacity (FVC) measured in liters (L).
Oscillometry | Screening, Day 1 and 28.
  Resistance measured in cm H2O s/L .
Oscillometry | Screening, Day 1 and 28.
  Resistance change measured in cm H2O s/L..
Oscillometry | Screening, Day 1 and 28.
  Reactance of respiratory system measured in cm H2O s/L.
Plethysmograhy | Screening and Day 28.
  Functional Residual Capacity (FRC) measured in liters (L).
Plethysmograhy | Screening and Day 28.
  Total Lung Capacity (TLC) measured in liters (L).
Plethysmograhy | Screening and Day 28.
  Ratio of Residual Volume measured as a percentage (%).
Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) | Screening and Day 28.
  DLCO measured in milliliters per min per millimeter of Mercury (mL/min/mmHg).
Pulse oximetry | Screening, Day 1, 2, 3, 4, 5, 8, 9, 21 and 28.
  Measuring oxygen saturation in the participants blood (SpO2)
6-minute walk-test | Screening, Day 1, 5, 9, 21 and 28.
  Assessment of exercise tolerance , distance walked in 6-minutes measured in meters (m).
Exhaled Nitirc Oxide Test | Screening, Day 1, 2, 3, 4, 5, 8, 9, 21 and 28.
  The fractional exhaled nitric oxide (FENO) test measures the amount of nitric oxide that is exhaled from a breath. It is a marker of lung inflammation, and is useful for differentiating asthma from COPD and other conditions presenting with similar symptoms [26]. FENO values of < 25 parts per billion (ppb) are considered normal, 25-50 ppb as intermediate and > 50 ppb as high.
St George Respiratory Questionnaire for COPD | Screening, Day 1, Day 28, Month 3 and Month 6.
  Measurement of quality of life validated for participants with COPD. Each subscale and the total score range from 0 (no impact) to 100 (worst possible impact).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wolf, Medical Doctor, Principal Investigator — Veritus Research
Locations (2):
- Australia (2):
  - Veritus Research, Bayswater, Victoria
  - Doherty Clinical Trials Limited, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
De-identified data will be published in a peer review scientific journal or presented at a scientific conference. There is no plan at this stage to make IPD available.